CLINICAL TRIAL: NCT01605292
Title: Radial Artery Access With Ultrasound Trial
Acronym: RAUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Lenox Hill Hospital (Other); Jamaica Hospital Medical Center (Other); Oklahoma City VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arnold Seto, Assistant Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-8432
Record Dates: First submitted 2012-01-26; First posted 2012-05-24 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Artery Disease
Keywords: Transradial catheterization; Ultrasound; Radial artery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpation (Active Comparator): Manual palpation of radial pulse, as sole guide to needle cannulation.
  Interventions: Procedure: Palpation
- Ultrasound (Experimental): Real-time ultrasound guidance to facilitate needle cannulation of artery.
  Interventions: Procedure: Ultrasound guidance

INTERVENTIONS:
Procedure: Ultrasound guidance — Real time ultrasound guidance using ultrasound probe covered in sterile plastic, visualizing radial artery while needle passage attempted.
  Arms: Ultrasound
Procedure: Palpation — Manual palpation for localizing radial artery for inserting needle.
  Arms: Palpation

SUMMARY:
Radial artery access for cardiac catheterization can require multiple attempts. Multiple attempts increase the time required, patient discomfort, and the risk of arterial spasm. Ultrasound guidance has been shown in other studies to reduce the number of attempts and complications in central venous and femoral artery access. This study will test if the addition of ultrasound guidance reduces the number of attempts and time required to access the radial artery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting for cardiac or peripheral catheterization with planned radial approach.
* Barbeau's or Allen's test indicating at least some degree of collateral circulation in palmar vessels
* Functional ultrasound equipment with ultrasound trained attending operator

Exclusion Criteria:

* Inability to provide informed consent
* Femoral access
* Emergency procedure (Shock, STEMI)
* End-stage renal disease on hemodialysis
* Previous ipsilateral puncture within 1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold H Seto, MD, MPA, Principal Investigator — University of California, Irvine and Long Beach VA Medical Center; Zoran Lasic, MD, Principal Investigator — Lenox Hill Hospital
Locations (6):
- United States (6):
  - Long Beach VA Medical Center, Long Beach, California
  - University of California Irvine Medical Center, Orange, California
  - Baptist Hospital of Miami, Miami, Florida
  - Jamaica Hospital, Jamaica, New York
  - Lenox Hill Hospital, New York, New York
  - Oklahoma VA Medical Center, Oklahoma City, Oklahoma

REFERENCES:
- [Result] Seto AH, Roberts JS, Abu-Fadel MS, Czak SJ, Latif F, Jain SP, Raza JA, Mangla A, Panagopoulos G, Patel PM, Kern MJ, Lasic Z. Real-time ultrasound guidance facilitates transradial access: RAUST (Radial Artery access with Ultrasound Trial). JACC Cardiovasc Interv. 2015 Feb;8(2):283-291. doi: 10.1016/j.jcin.2014.05.036. Epub 2015 Jan 14. PMID 25596790
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palpation | Ultrasound
Started | 351 | 347
Completed | 351 | 347
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palpation | Ultrasound | Total
Number analyzed (Participants) | 351 | 347 | 698
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.6) | 61.5 (11.5) | 61.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 93 | 182
  Male | 262 | 254 | 516
Outpatient [Number; unit: participants]
  Outpatient | 141 | 139 | 280
  Inpatient or admitted | 210 | 208 | 418
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (7.2) | 30.4 (6.9) | 30.3 (7.0)
Obesity, BMI >= 30 [Number; unit: participants]
  Obese | 153 | 149 | 302
  Nonobese | 198 | 198 | 396
Hypertension [Number; unit: participants]
  HTN | 305 | 292 | 597
  Non-HTN | 46 | 55 | 101
Hypercholesterolemia [Number; unit: participants]
  Hypercholesterolemia | 265 | 254 | 519
  Normal cholesterol | 86 | 93 | 179
Diabetes mellitus [Number; unit: participants]
  DM | 151 | 149 | 300
  No DM | 200 | 198 | 398
Tobacco [Number; unit: participants]
  Tobacco use | 107 | 128 | 235
  No tobacco use | 244 | 219 | 463
Peripheral vascular disease [Number; unit: participants]
  PVD | 16 | 14 | 30
  No PVD | 335 | 333 | 668
Barbeau class B or C [Number; unit: participants] — Of those patients receiving Barbeau's test. Barbeau's Class A reflects no reduction of arterial waveform on pulse oximetry after radial artery occlusion, indicating robust collateral flow from the ulnar artery. Barbeau's Class B and C reflect delayed but eventual recovery of arterial waveform on pulse oximetry after radial artery occlusion, indicating the presence of some but limited collaterals from the ulnar artery. Barbeau's Class D patients (no demonstrable collaterals) were excluded from the study.
  participants
    Barbeau's Class A | 95 | 93 | 188
    Barbeau's Class B or C | 54 | 56 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Attempts
Description: Number of passes of the needle required to access the artery during the cardiac catheterization procedure. This is only assessed at the time of the procedure, i.e. during the first 30 minutes. This is to be reported as both total number of attempts and as a first pass success rate.
Time Frame: Immediately during procedure. (up to 30 minutes)
Population: 473 patients of 698 had number of attempts measured correctly by number of forward passes. This subgroup of the whole population was used for analysis of number of attempts.
Measure: Mean (Standard Deviation); unit: forward attempts
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 237 | 236
forward attempts | 3.05 (3.4) | 1.65 (1.2)
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Time to Sheath Insertion (Seconds)
Description: Time from initiation of vascular access attempts to successful aspiration or flushing of the sheath. Time for lidocaine administration, palpation of pulse, or imaging is excluded.
Time Frame: Immediately during procedure (within 30 minutes)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 351 | 347
seconds | 108 (112) | 88 (78)
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p = 0.006, t-test, 2 sided

3. Secondary Outcome: First-pass Success Rate
Description: Proportion of procedures achieving access on the first attempt
Time Frame: Immediate
Population: Subgroup of patients with accurate number of attempts measured
Measure: Number; unit: participants
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 237 | 236
participants
  Successful first-pass | 104 | 153
  Unsuccessful first-pass | 133 | 83
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Other Pre Specified Outcome: Radial Artery Spasm
Description: Spasm defined and identified by the operator as any significant resistance or patient pain with catheter manipulation
Time Frame: Immediately during procedure (within 30 min)
Measure: Number; unit: participants
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 351 | 347
participants | 12 | 15
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p = 0.56, Fisher Exact

5. Other Pre Specified Outcome: Difficult Access Procedures >= 5 Attempts
Description: Difficult procedures were defined as either requiring >= 5 attempts
Time Frame: Immediately during procedure (within 30 min)
Measure: Number; unit: participants
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 237 | 236
participants
  >=5 attempts | 44 | 6
  <5 attempts | 193 | 230
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p < 0.0001, Fisher Exact

6. Other Pre Specified Outcome: Difficult Access >= 5 Minutes
Description: Access that requires >= 5 minutes from first attempt to sheath insertion
Time Frame: Immediate (within 30 minutes)
Measure: Number; unit: participants
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 351 | 347
participants
  >= 5 minutes | 24 | 13
  < 5 minutes | 327 | 334
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p = 0.07, Chi-squared

7. Other Pre Specified Outcome: Bleeding Complication
Description: Any hematoma >2 cm or bleeding requiring intervention
Time Frame: After procedure (within 24 hours)
Measure: Number; unit: participants
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 351 | 347
participants | 4 | 5
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p = 0.75, Fisher Exact

8. Post Hoc Outcome: Crossover to Ultrasound Rescue Attempts After 5 Minutes
Description: Patients randomized to palpation-guided access could have their procedure changed to ultrasound at operator discretion after 5 minutes of palpation-guided attempts.
Time Frame: 5 minutes
Population: Only patients randomized to palpation could potentially cross over to ultrasound technique.
Measure: Number; unit: participants
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 10 | 0
participants
  Successful rescue with ultrasound | 8 |
  Unsuccessful rescue with ultrasound | 2 |

9. Post Hoc Outcome: Failure of Radial Sheath Insertion With Original Randomized Technique
Time Frame: Immediate
Measure: Number; unit: participants
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 351 | 347
participants | 15 | 3
Statistical Analysis 1: Comparison: Palpation vs Ultrasound; Test type: Superiority or Other; p = 0.007, Fisher Exact

10. Other Pre Specified Outcome: Pain Score
Description: Patient-reported wrist pain using a visual-analogue scale (0-10) 2-8 hours after the procedure, where 0 is no pain and 10 is severe pain.
Time Frame: 2-8 hours after procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Palpation | Ultrasound
Number analyzed (Participants) | 351 | 347
units on a scale | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Arm/Group | Palpation | Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/351 | 0/347
Other Adverse Events (participants affected / at risk) | 0/351 | 0/347

LIMITATIONS AND CAVEATS:
Blinding was not possible in this study. We cannot exclude a bias in the performance, measurement, or recording of the procedure or clinical data. Time to prepare the US probe was not included in the time to access.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No